CLINICAL TRIAL: NCT05575752
Title: Acute Health Effects of High Temperature Exposure in Healthy Young Adults: a Randomized Controlled Study
Brief Title: Acute Health Effects of High Temperature Exposure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haidong Kan, Professor, Fudan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FDUEH-8
Record Dates: First submitted 2022-09-28; First posted 2022-10-12 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular System; Respiratory System; Cognitive Function
Keywords: High Temperature; Randomized controlled trial; Cardiovascular effects; cognitive function
MeSH Terms: conditions — Fever | interventions — Diathermy; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high temperature (32℃) group (Experimental): Subjects in exposure group will be exposed to high temperature (32℃) for about 2 hours in a chamber.
  Interventions: Other: high temperature (32℃) group
- moderate temperature (22℃) group (Sham Comparator): Subjects in exposure group will be exposed to moderate temperature (22℃) for about 2 hours in a chamber.
  Interventions: Other: moderate temperature (22℃) group

INTERVENTIONS:
Other: high temperature (32℃) group — The exposure group will be exposed to high temperature (32℃) in a chamber for about 2 hours, resting during the whole periods.
  Arms: high temperature (32℃) group
Other: moderate temperature (22℃) group — The exposure group will be exposed to thermoneutral temperature (22℃) in a chamber for about 2 hours, resting during the whole periods.
  Arms: moderate temperature (22℃) group

SUMMARY:
This is a randomized controlled human exposure crossover study. Investigators aims to assess the acute effects of high temperature exposure and the underlying mechanisms.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled human exposure crossover study among about 30 healthy young adults in Shanghai, China. Each subject will be exposed twice: once to the high temperature (32℃) and once to moderate temperature (22℃) in a chamber for about 2 hours. During the exposure session, each subject will be requested to rest. Health examinations will be conducted immediately prior to exposure, during the period of exposure and after exposure. Health examinations include symptom questionnaire, blood pressure tests, cognitive function tests, magnetic resonance imaging, skin tests, spirometry, and Holter monitoring. Investigators plan to collect blood, urine and oropharyngeal swabs samples.

ELIGIBILITY:
Inclusion Criteria:

* Living in Shanghai during the study period;
* Body mass index > 18.5 and ≤ 28;
* right-handed;
* receiving or having received higher education;
* with ability to read and understand Chinese smoothly.

Exclusion Criteria:

* Smoking and alcohol abuse;
* Current drug and dietary supplements intake;
* Subjects with allergic diseases, such as allergic rhinitis, allergic asthma, and atopy;
* Subjects with cardiovascular diseases, such as congenital heart disease, pulmonary heart disease, and hypertension;
* Subjects with respiratory diseases, such as asthma, chronic bronchitis, and chronic obstructive pulmonary disease;
* Subjects with chronic diseases, such as diabetes, chronic hepatitis, and kidney disease;
* Subjects who have a history of major surgery due to the cardiovascular, cerebrovascular, respiratory, or neurological diseases;
* Subjects with neurologic disorders, such as stroke, traumatic brain injury, epilepsy, and schizophrenia;
* Abnormal spirometry (FEV1 and FVC ≤ 75% of predicted and FEV1/FVC ≤ 0.65);
* Subjects with color vision disabilities.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-23 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of pulse wave velocity measured by an arteriography device performing oscillometric measurement | Pulse wave velocity will be examined before exposure and immediately after the exposure session
  Pulse wave velocity (PWV) is one of the arterial stiffness indicators. The changes of PWV will be measured.
Changes of AIx@75 measured by an arteriography device performing oscillometric measurement | AIx@75 will be examined before exposure and immediately after the exposure session
  Augmentation index normalized to 75 bpm heart rate (AIx@75) is one of the arterial stiffness indicators. The changes of AIx@75 will be measured.
Changes of reflection magnitude measured by an arteriography device performing oscillometric measurement | Reflection magnitude will be examined before exposure and immediately after the exposure session
  Reflection magnitude is one of the arterial stiffness indicators. The changes of reflection magnitude will be measured.
Results of Stroop Tests | The tests will be conducted before exposure and immediately after the exposure session
  Investigators plan to measure the changes of cognitive function using Stroop Test. The time taken to complete the test could reflect cognitive function, and a shorter time means better cognitive function.
Changes of forced expiratory volume in the first second (FEV1) | The tests will be examined before exposure and half an hour after exposure
  Investigators plan to measure the changes of the forced expiratory volume in 1 s (FEV1) using a smart spirometer (Model A1, BreathHome, China) supervised by professional medical staff. Before the pulmonary function test, subjects will practice several times by themselves. During the examination, each subject stands and clamps the nose clip, and repeats the test, with the best result as the criterion. FEV1 reflect pulmonary function.
Changes of forced vital capacity (FVC) | FVC will be examined before exposure and half an hour after exposure
  Investigators plan to measure the changes of forced vital capacity (FVC) using spirometer (Model A1, BreathHome, China). FVC reflects the expiratory resistance of large airways.
Changes of peak expiratory flow rate (PEF) | FVC will be examined before exposure and half an hour after exposure
  Investigators plan to measure the changes of peak expiratory flow (PEF) using smart spirometer (Model A1, BreathHome, China). PEF reflects airway patency and respiratory muscle strength.
Changes of maximum expiratory flow rate at 25% vital capacity (MEF25) | MEF25 will be examined before exposure and half an hour after exposure
  Investigators plan to measure the changes of maximum expiratory flow rate at 25% vital capacity. MEF25% reflects the early stage of expiratory flow rate.
Changes of maximum expiratory flow rate at 50% vital capacity (MEF50) | MEF50 will be examined before exposure and half an hour after exposure
  Investigators plan to measure the changes of maximum expiratory flow rate at 50% vital capacity using smart spirometer (Model A1, BreathHome, China). MEF50 reflects the interim stage of expiratory flow rate.
Changes of maximum expiratory flow rate at 75% vital capacity (MEF75) | MEF75 will be examined before exposure and half an hour after exposure
  Investigators plan to measure the changes of maximum expiratory flow rate at 50% vital capacity (MEF75%) using smart spirometer (Model A1, BreathHome, China). MEF75 reflects the terminal stage of expiratory flow rate.

SECONDARY OUTCOMES:
Blood Pressure | Blood pressure will be examined before exposure and immediately after the exposure session
  The changes of systolic blood pressure (SBP) and diastolic blood pressure (DBP) will be measured.
Results of Schulte table Tests | The tests will be conducted before exposure and immediately after the exposure session
  Investigators plan to measure the changes of cognitive function using Schulte table. The time taken to complete the test and the accuracy could reflect cognitive function. Less time and greater accuracy mean better cognitive function.
Activated brain regions demonstrating neural activity related to the high temperature exposure | 1 hour after exposure session
  Investigators plan to measure brain activity associated with high temperature exposure by magnetic resonance imaging (MRI). Brain imaging data will be extracted from MRI data. The fractional amplitude of low frequency fluctuation (fALFF) would be extracted to reflect neural activity of brain regions.
Activated brain regions demonstrating neural connectivity related to the high temperature exposure | 1 hour after exposure session
  Investigators plan to measure brain activity associated with high temperature exposure by magnetic resonance imaging (MRI). Brain imaging data will be extracted from MRI data. The degree of centrality (DC) would be extracted to reflect neural connectivity of brain regions.
Activated brain regions demonstrating neural synchronization related to the high temperature exposure | 1 hour after exposure session
  Investigators plan to measure brain activity associated with high temperature exposure by magnetic resonance imaging (MRI). Brain imaging data will be extracted from MRI data. The regional homogeneity (ReHo) would be extracted to reflect neural synchronization of brain regions.
Changes of airway inflammation indicator fractional concentration of carbon monoxide (FeCO) | FeCO will be examined before exposure and half an hour after exposure
  Investigators plan to measure the changes of fractional concentration of carbon monoxide.
Changes of airway inflammation indicator fractional exhaled nitric oxide (FeNO) | FeNO will be examined before exposure and half an hour after exposure
  Investigators plan to measure the changes of fractional exhaled nitric oxide.

OTHER OUTCOMES:
Changes of the scores of thermal sensation questionnaires | before exposure and immediately after the exposure session
  Changes of scores of thermal sensation questionnaires which ranged from -5 to 5. Zero score refers to the thermal comfort sensation. Higher scores refer to more uncomfortable sensations of hot. Lower scores refer to more uncomfortable sensations of cold.
Differences in RNA expression levels detected in serum transcriptomics between the two exposures | 1 hour after the exposure session
  Illumina-based transcriptomics is non-targeted. The study is to find the differentially expressed exosome RNA in serum after high temperature exposure
Differences in protein levels detected in blood Clara cell protein (CC16) between the two exposures | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Investigators plan to measure the changes of Clara cell protein using enzyme linked immunosorbent assay (ELISA). Clara cell protein (CC16) indicate lung epithelial injury.
Differences in protein levels detected in blood chitinase-3-like protein 1 (YKL-40) between the two exposures | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Investigators plan to measure the changes of chitinase-3-like protein 1 protein using enzyme linked immunosorbent assay (ELISA). YKL-40 represents airway inflammation and remodeling.
Changes of heart rate variability (HRV) parameter RMSSD | Volunteers will be asked to wear electrographic Holter monitors for 24 hours from 1:00 P.M. at the day of intervention to 1:00 P.M. at the next day.
  Investigators plan to measure the changes of HRV parameter the root mean square of successive differences between adjacent normal cycles (RMSSD) .
Changes of heart rate variability (HRV) parameter SDNN | Volunteers will be asked to wear electrographic Holter monitors for 24 hours from 1:00 P.M. at the day of intervention to 1:00 P.M. at the next day.
  Investigators plan to measure the changes of heart rate variability parameter standard deviation of NN intervals (SDNN) .
Changes of heart rate variability (HRV) parameter PNN50 | Volunteers will be asked to wear electrographic Holter monitors for 24 hours from 1:00 P.M. at the day of intervention to 1:00 P.M. at the next day.
  Investigators plan to measure the changes of heart rate variability parameter percent of NN50 in the total number of NN intervals (PNN50).
Differences in metabolic profiling detected in blood between the two exposures | 1 hour after the exposure session
  The differential metabolic profiling in blood related to high temperature exposure will be detected by mass spectrometry-based non-targeted metabolomics.
Differences in protein levels detected in blood between the two exposures | 1 hour after the exposure session
  The differentially expressed proteins in blood related to high temperature exposure will be detected by non-targeted proteomics.
Differences in DNA methylation levels detected in whole-blood between the two exposures | 1 hour after the exposure session
  Genome-wide DNA methylation in whole-blood were detected using Illumina 935K Beadchip. The study is to identify differential CpG loci after high temperature exposure.
Change in tumor necrosis factor-α (TNF-α) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of TNF-α in blood.
Change in C reactive protein (CRP) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of C reactive protein in blood.
Change in oxidized low density lipoprotein (Ox-LDL) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of Ox-LDL in blood.
Change in malondialdehyde (MDA) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of MDA in blood.
Change in von Willebrand factor (vWF) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of vWF in blood.
Change in fibrinogen concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of fibrinogen in blood.
Change in endothelial nitric oxide synthase (eNOS) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of eNOS in blood.
Change in endothelin-1 (ET-1) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of ET-1 in blood.
Change in blood glucose concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of blood glucose.
Change in insulin concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of insulin in blood.
Change in low-density lipoprotein cholesterol (LDL) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of LDL in blood.
Change in total cholesterol (TC) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of TC in blood.
Change in apolipoprotein B (ApoB) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of ApoB in blood.
Change in matrix metallopeptidase 2 (MMP2) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of MMP2 in blood.
Change in matrix metallopeptidase 9 (MMP9) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of MMP9 in blood.
Changes of skin sebum level | 60 minutes and 120 minutes of exposure.
  Evaluation of the differential sebum level between the two groups
Changes of facial secreted sebum composition | One hour after the exposure session
  Evaluation of the differential facial secreted sebum composition between the two groups
Changes of the luminosity on the cheeks | before exposure and at 40 minutes after the end of exposure
  Evaluation of the differential facial luminosity between the two groups. The luminosity on the cheeks of the participants were visually assessed by the dermatologist with the naked eyes. The skin luminosity was rated on a 4-point scale (0 to 3, with larger scores indicating more glossy).
Changes of the pores on the cheeks | before exposure and at 40 minutes after the end of exposure
  Evaluation of the differential pores sizes between the two groups. The pores on the cheeks of the participants were visually assessed by the dermatologist with the naked eyes. The pore appearance was rated on a 6-point scale (0 to 5, with larger scores indicating larger pore size).
Changes of subjective skin sensations | 30, 60, 90, and 120 minutes after the start of each exposure session
  Evaluation of the differential subjective skin sensations between the two groups. The questionnaire consisted of seven questions regarding dryness, oiliness, stickiness, tightening, itchiness, tingling, and freshness. Each participant was asked to self-evaluate their skin sensations on a 4-point scale from 0 to 3, indicating "not at all", "somewhat", "fairly", and "fully compliant".
Changes of stratum corneum protein levels | within 30 minutes after the end of exposure
  Evaluation of the differential stratum corneum (SC) protein levels between the two groups
Differences in lipid metabolites levels detected in skin surface between the two exposures | Skin surface sebum was collected 5 minutes after exposure
  The differentially lipid metabolites levels in skin surface related to high temperature exposure will be detected by targeted quantitative lipidomic analysis.
Change in total antioxidant capacity of collected stratum corneum | within 30 minutes after the end of exposure
  Change of the total antioxidant capacity in collected stratum corneum will be measured.
Change in kallikrein-5 concentrations of collected stratum corneum | within 30 minutes after the end of exposure
  Change of the concentrations of kallikrein-5 in collected stratum corneum will be measured.
Change in interleukin-1α concentrations of collected stratum corneum | within 30 minutes after the end of exposure
  Change of the concentrations of interleukin-1α in collected stratum corneum will be measured.
Change in total protein concentrations of collected stratum corneum | within 30 minutes after the end of exposure
  Change of the concentrations of total protein in collected stratum corneum will be measured.
Change in interleukin-1 receptor antagonist concentrations of collected stratum corneum | within 30 minutes after the end of exposure
  Change of the concentrations interleukin-1 receptor antagonist in collected stratum corneum will be measured.
Differences in protein levels related to cardiovascular system and inflammation detected in blood between the two exposures | 1 hour after the exposure session
  The differentially expressed proteins in blood related to cardiovascular system and inflammation after high temperature exposure will be detected by targeted Olink proteomics.
Change in brain-derived neurotrophic factor (BDNF) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of BDNF in blood.
Change in glial cell line-derived neurotrophic factor (GDNF) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of GDNF in blood.
Change in Gamma-aminobutyric acid (GABA) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of GABA in blood.
Change in glutathione (GSH) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of IFN in blood.
Change in interferon (IFN) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of IFN in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Kan, PhD, Study Director — Department of Environmental Health, School of Public Health, Fudan University
Locations (1):
- Department of Environmental Health, School of Public Health, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT05575752/SAP_000.pdf